CLINICAL TRIAL: NCT05683470
Title: Expanded Access to RBS2418 for an Individual Patient With Pancreatic Cancer
Brief Title: Expanded Access RBS2418 Treatment
Status: No longer available | Type: Expanded Access
Sponsor: Riboscience, LLC. (Industry)
Collaborators: Dr. Bertrand Tuan (Unknown)
Responsible Party: Sponsor
Other Study IDs: RBS2418-EA-002
Record Dates: First submitted 2022-12-26; First posted 2023-01-13 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Expanded Access in Pancreatic Cancer

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: RBS2418 — RBS2418 will be administered orally at 200 mg two times per day (BID).

SUMMARY:
This is an expanded access treatment protocol designed to provide access of RBS2418 to a single patient with pancreatic cancer.

DETAILED DESCRIPTION:
Given lack of any therapeutic options such as standard of care chemotherapy for this single patient owing to lack of tolerability and opportunity to enroll in any clinical trial due to extent of disease, patient desires to try compassionate use protocol with RBS2418, an oral immunotherapeutic agent that is currently in clinical trials and is well tolerated by patients. Furthermore, patient's tumor has been shown to express ENPP1, the protein targeted by RBS2418

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and able to provide informed consent. Only the patient for whom this clinical study/experimental treatment was designed will be given the investigational drug under the treatment of the PI. No other patient is authorized to participate in or to receive treatment under this treatment protocol.

Exclusion Criteria:

* Not applicable

Sex: Female
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Tuan, MD, Principal Investigator — Pacific Hematology and Oncology Associates